CLINICAL TRIAL: NCT01209377
Title: Randomized Controlled Study of Eye Movement Desensitization and Reprocessing (EMDR) Working Mechanism
Brief Title: Study of Eye Movement Desensitization and Reprocessing (EMDR) Working Mechanism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: German Research Foundation (Other); University of Giessen (Other)
Responsible Party: Martin Sack, MD, Technical University of Munich
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SA1475/2-1
Record Dates: First submitted 2010-06-17; First posted 2010-09-27 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: standard; fixed; no focus; EMDR treatment with bilateral stimulation via eye movement; EMDR treatment with fixed eyes; Trauma exposition without external stimulus
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard (Experimental): EMDR treatment with bilateral stimulation via eye movement
  Interventions: Behavioral: standard; Procedure: EMDR
- fixed (Experimental): EMDR treatment with eyes fixed
  Interventions: Behavioral: fixed; Procedure: EMDR
- no focus (Experimental): trauma exposition without external stimulus
  Interventions: Behavioral: no focus; Procedure: EMDR

INTERVENTIONS:
Behavioral: standard — EMDR treatment with bilateral stimulation via eye movement
  Arms: standard
Behavioral: fixed — EMDR treatment with fixed eyes
  Arms: fixed
Behavioral: no focus — trauma exposure without external focus
  Arms: no focus
Procedure: EMDR — Eye Movement Desensitization and Reprocessing (EMDR)

SUMMARY:
EMDR (Eye Movement Desensitization and Reprocessing) is an exposure-based procedure for the treatment of patients with post-traumatic stress disorder (PTSD). Although the efficiency of EMDR-treatment is empirically proven, it remains unclear whether the bilateral stimulation triggered via eye movements has specific effects on treatment outcome. Hypothesis explaining the efficacy of the EMDR treatment are: focussing on the moving hand triggers an orientation reaction, and the duality of alertness focus during trauma exposition causes a distraction of the traumatic topic.

Within a randomized controlled study 120 patients will be treated during 8 therapeutical sessions with EMDR with bilateral stimulation or one of two control conditions: EMDR without bilateral stimulation (eyes on a fixed, unmoving hand) and exposition without any visual stimuli to focus attention on. Primary outcome are scores on an interview measure for PTSD symptoms (Clinician Administered PTSD Scale (CAPS))as assessed pre-treatment and after treatment (max 8 sessions of psychotherapy).

The following hypothesis are investigated in the study:

1. EMDR treatment with bilateral stimulation through eye movements will be followed significant larger reduction in CAPS compared with EMDR treatment without bilateral stimulation (specific treatment effect of eye movements)
2. EMDR with eyes fixed will be followed by a significant larger reduction in CAPS compared with EMDR without external focus (specific treatment effect of distraction)

ELIGIBILITY:
Inclusion Criteria:

* the participant is able to reduce stress symptoms
* no actual contact to offender

Exclusion Criteria:

* drug or alcohol addiction
* inability to tell about the traumatic events
* cardiac problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-01 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
CAPS-2: Clinical Administered PTSD Scale | 30 minutes

SECONDARY OUTCOMES:
IES - Impact of Events Scale | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sack, PHD, Study Director — Technical University of Munich
Locations (1):
- Technische Universität München, Munich, Germany, Germany